CLINICAL TRIAL: NCT06079255
Title: Early Ischemia Detection by a Tissue CO2-sensor During Development of Acute Compartment Syndrome
Brief Title: Ischemia Detection During Development of Acute Compartment Syndrome
Acronym: IDEA
Status: Not yet recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sensocure AS (Industry)
Responsible Party: Principal Investigator, John Clarke-Jenssen, Chief Consultant, Oslo University Hospital
Other Study IDs: IDEA
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Ischemia Limb; Blood Circulation Disorder; Carbon Dioxide; Biosensing Techniques; Compartment Syndrome of Leg
Keywords: Ischemia; Biosensor; Carbon dioxide; Orthopedic surgery; Limb; Acute compartment syndrome
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IscAlert sensor in patient with risk of acute compartment syndrome: Patients admitted with leg injury at risk of acute compartment syndrome will receive IscAlert sensor(s) in the anterior compartment of the lower limb. A duration of maximum 10 days.
  Interventions: Device: IscAlert sensor(s) in patient with risk of acute compartment syndrome

INTERVENTIONS:
Device: IscAlert sensor(s) in patient with risk of acute compartment syndrome — of the replanted extremity Insertion of a CO2- and temperature sensor(s) (IscAlert) in the anterior compartment of a lower limb (leg)

SUMMARY:
This is an open, observational, prospective, descriptive, single-centre study including 60 patients. The study is designed to investigate if IscAlert sensor system can be used for reliable and continuous tissue carbon dioxide (pCO2)- and temperature monitoring in muscular tissue in lower extremity in patients at risk of developing acute compartment syndrome.

DETAILED DESCRIPTION:
This is an open, observational, prospective, descriptive, single-centre study including 60 patients. The study is designed to investigate if IscAlert sensor system can be used for reliable and continuous tissue carbon dioxide (pCO2)- and temperature monitoring in muscular tissue in lower extremity in patients at risk of developing acute compartment syndrome.

The study will provide information regarding the clinical usefulness of tissue perfusion assessment by pCO2 and temperature monitoring in the diagnosis of patients at risk of developing acute compartment syndrome. Additionally, it will provide information regarding limits of pCO2 and temperature in the tissue indicating the need for fasciotomy. A fasciotomy will be performed independent of the measured pCO2 and temperature measurements in the muscle if clinical signs indicate a development of possible acute compartment syndrome. Measures of pain, and number of infections and bleeding caused by (or assumed to be caused by IscAlert) at insertion site will be registered.

The duration of investigation: In a patient: From insertion of first IscAlert™ sensor(s) to discharge from hospital. The sensors will usually be implanted for two days each. Follow up until 30 days after discharge from the hospital. 13 months of inclusion of all patients. There will be one last follow-up visit 1 year after discharge which will only look at sequelae after acute compartment syndrome and not sensors related issues.

Primary Aim: To assess if pCO2-levels when assessed with IscAlert correctly indicate the presence of acute compartment syndrome in muscular tissue in lower extremity in patients at risk of developing acute compartment syndrome.

Hypotheses

1. The pCO2 measurements will be at least 3 kPa higher when assessed with IscAlert in the muscle compartment where acute compartment syndrome develops compared to compartments where acute compartment syndrome does not develop.
2. No clinically significant pain, bleeding or infection will occur due to using IscAlert.
3. The temperature measurements will be lower when assessed with IscAlert in the muscle compartment where acute compartment syndrome develops compared to compartments where acute compartment syndrome does not develop.

ELIGIBILITY:
Inclusion Criteria:

* Must have a leg fracture that, perceived by the clinician, could give rise to later developing acute compartment syndrome condition.
* Subject must be 18 years or more.
* Able to sign informed consent.
* Expected cooperation of the patients for the treatment and follow up

Exclusion Criteria:

* Another study interfering with current study
* Any reason why, in the opinion of the investigator, the patient should not participate.
* Patients where a fasciotomy has already been decided should be performed

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 consecutive patients at risk of acute compartment syndrome of both genders at the age above 18 years who corresponds to inclusion and exclusion criteria at Oslo University Hospital will be included
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Tissue CO2-level | 10 days
  Tissue CO2-level (kPa) during insertion period

SECONDARY OUTCOMES:
Bleeding | 10 days
  Amount of blood from insertion site (ml)
Infection | 30 days
  Infection from insertion site at the discretion of the investigator (yes or no)
Pain at sensor insertion site | 30 days
  Pain at the insertion site measured by Numeric Rating Scale (0= no pain, 10= maximum pain)
Pain in the lower leg during hospitalisation | 10 days
  Pain in the injured lower leg measured by Numeric Rating Scale (0= no pain, 10= maximum pain)
Color of the lower leg | 10 days
  Skin color of the injured lower leg (Blue/Pink/Pale/Normal) during hospitalisation
Paresthesia of the lower leg | 10 days
  Paresthesia of the injured lower leg (Yes/No) during hospitalisation
Paralysis of the lower leg | 10 days
  Paralysis of the injured lower leg (Yes/No) during hospitalisation
Lenght of sensor implantation time | 10 days
  Lenght of sensor implantation time during hospitalisation
Time to discovery of reduced blood flow in lower leg | 10 days
  Number of days and hours from primary surgery end to obstructed blood flow is diagnosed.
Number of re-operations | 30 days
  Number of reoperations (fasciotomies) caused by acute compartment syndrome
Number of skin grafts performed | 1 year
  Number of skin grafts performed caused by sequelae after acute compartment syndrome
Number of limb amputations performed | 1 year
  Number of limb amputations performed caused by sequelae after acute compartment syndrome
Number of sensory deficit conditions | 1 year
  Number of sensory deficit conditions caused by sequelae after acute compartment syndrome
Number of paralysis conditions | 1 year
  Number of paralysis conditions caused by sequelae after acute compartment syndrome
Number of rhabdomyolysis conditions | 1 year
  Number of rhabdomyolysis conditions caused by sequelae after acute compartment syndrome
Number of limb muscle contractures | 1 year
  Number of limb muscle contractures caused by sequelae after acute compartment syndrome
Number of acute compartment syndrome conditions during hospitalisation | 30 days
  Number of acute compartment syndrome conditions during hospitalisation
Number of acute compartment syndrome conditions after 1 year | 1 year
  Number of acute compartment syndrome conditions after 1 year
Incidence of death 1 year | 1 year
  Mortality 1 year after admission
Incidence of death during hospitalisation | 30 days
  Mortality during primary hospitalisation
Lenght of stay during primary hospitalisation | 30 days
  Lenght of stay during primary hospitalisation
Number of pack-years | 30 days
  Smoking habit; number of pack-years by participants
Intravenous fluid | 12 hours
  Intravenous fluid given during surgery (ml)
Vasoactive drugs | 12 hours
  Vasoactive drugs given during surgery (microgram)
Tissue temperature level | 10 days
  Tissue temperature level (grade Celcius) during insertion period
IscAlert functionality | 10 days
  Number of hours with a well-functioning sensor (giving CO2- and temperature data)
Intracompartmental pressure | 10 days
  Intracompartmental pressure (mmHg) measured in anterior compartment of the injured leg
Systolic blood pressure during hospitalisation | 10 days
  Systolic blood pressure (mmHg) during hospitalisation
Diastolic blood pressure during hospitalisation | 10 days
  Diastolic blood pressure (mmHg) during hospitalisation
Peripheral pulse during hospitalisation | 10 days
  Peripheral distal pulse (rate/minute) at the injured leg during hospitalisation
Hemoglobin | 10 days
  Hemoglobin (g/dL) level during hospitalisation
Creatine kinase | 10 days
  Creatine kinase (U/L) level during hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: John Clarke-Jenssen, MD, PhD., Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD to other researchers